CLINICAL TRIAL: NCT04722848
Title: Newly Diagnosed Adult Philadelphia Chromosome-Positive Acute Lymphoblastic Leukemia (Ph+ ALL). Sequential Treatment With Ponatinib and the Bispecific Monoclonal Antibody Blinatumomab vs Chemotherapy and Imatinib
Brief Title: Sequential Treatment With Ponatinib and Blinatumomab vs Chemotherapy and Imatinib in Newly Diagnosed Adult Ph+ ALL
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALL2820
Record Dates: First submitted 2021-01-20; First posted 2021-01-25 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Acute Lymphoblastic Leukemia (Philadelphia Chromosome Positive); ALL, Adult; Philadelphia-Positive ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — ponatinib; blinatumomab; Drug Therapy; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ponatinib+Blinatumomab (Experimental): patients will receive induction with ponatinib followed by at least 2 cycles of blinatumomab
  Interventions: Drug: Ponatinib + Blinatumomab
- Chemotherapy+Imatinib (Active Comparator): patients will receive a combination of imatinib and chemotherapy.
  Interventions: Drug: Chemotherapy + Imatinib

INTERVENTIONS:
Drug: Ponatinib + Blinatumomab — Patients aged 18-65 will receive Ponatinib at the dose of 45 mg/day for the first 22 days and then will reduce the dose to 30 mg (depending on the morphologic and molecular response), whereas patients older than 65 years will start Ponatinib at 30 mg/day, in order to avoid TAEs. Patients will continue treatment with Ponatinib up to day 70 (10 weeks of treatment), except for disease progression, intolerable toxicity, or withdrawal from study. Thereafter:
  * Patients will receive Blinatumomab (minimum 2 cycles, up to a maximum of 5).
  * Patients not achieving a CHR after 2 cycles of Blinatumomab will go off-study. After the 2 cycles of Blinatumomab patients aged 18-65 will be stratified for transplant allocation
  Arms: Ponatinib+Blinatumomab
Drug: Chemotherapy + Imatinib — patients aged 18-65 will receive chemotherapeutic scheme combined with Imatinib. Elderly patients will receive Imatinib plus mild chemotherapy.
  Arms: Chemotherapy+Imatinib

SUMMARY:
This is a randomised, open-label, multicenter, phase III study for adult de novo Ph+ ALL patients based on the combination of Ponatinib with Blinatumomab. The control arm will be represented by a chemotherapeutic scheme combined with Imatinib for patients aged 18-65 and by Imatinib plus age-adjusted chemotherapy for elderly patients (>65 years old).

Patients will be randomized 2:1 to receive the experimental or control arm. If patients in the control arm do not achieve a CHR and/or MRD negativity, after the sixth consolidation cycle (week 20), a crossover to receive Blinatumomab is planned. Likewise, if patients in the control arm develop an ABL1 mutation at any time of treatment, they will switch to experimental arm. HLA typing will be performed immediately after diagnosis in both arms for patients aged up to 65 years.

After the 2 cycles of Blinatumomab in the experimental arm and after consolidation in the control arm, patients aged 18-65 will be stratified for transplant allocation.

DETAILED DESCRIPTION:
This is a randomised, open-label, multicenter, phase III study for adult de novo Ph+ ALL patients (≥18 years, no upper age-limit) based on the combination of the pan-TKI Ponatinib, with the bispecific monoclonal antibody Blinatumomab. The control arm will be represented by a chemotherapeutic scheme combined with Imatinib for patients aged 18-65 and by Imatinib plus age-adjusted chemotherapy for elderly patients (>65 years old).

Patients (≥18 years, no upper age limit) will be randomized 2:1 to receive the experimental or control arm. If patients in the control arm do not achieve a CHR and/or MRD negativity, after the sixth consolidation cycle (week 20), a crossover to receive Blinatumomab is planned. Likewise, if patients in the control arm develop an ABL1 mutation at any time of treatment, they will switch to experimental arm. HLA typing will be performed immediately after diagnosis in both arms for patients aged up to 65 years.

After the 2 cycles of Blinatumomab in the experimental arm and after consolidation in the control arm, patients aged 18-65 will be stratified for transplant allocation.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent according to ICH/EU/GCP and national local laws.
2. Newly diagnosed adult B-precursor Ph+ ALL patients.
3. WHO performance status less or equal to 2.
4. Age greater or equal to18 years, with no upper age limit.
5. Renal and hepatic function as defined below:

   * AST (GOT), ALT (GPT), and AP <2 x upper limit of normal (ULN).
   * Total bilirubin <1.5 x ULN.
   * Creatinine clearance equal or greater than 50 mL/min.
6. Pancreatic function as defined below:

   * Serum amylase less or equal to 1.5 x ULN and serum lipase less or equal to1.5 x ULN.
7. Normal cardiac function.
8. No evidence of CNS leukemia at blinatumomab start.
9. Negative HIV test, negative hepatitis B (HBsAg) and hepatitis C virus (anti-HCV) test.
10. Negative pregnancy test in women of childbearing potential.
11. Bone marrow specimen from primary diagnosis available.

Exclusion Criteria:

1. History of or current relevant CNS pathology (ongoing grade ≥2 epilepsy, seizure, paresis, aphasia, clinically relevant apoplexia, severe brain injuries, dementia, Parkinson's disease, organic brain syndrome, psychosis).
2. Impaired cardiac function, including any one of the following:

   * LVEF <45% as determined by MUGA scan or echocardiogram.
   * Complete left bundle branch block.
   * Use of a cardiac pacemaker.
   * ST depression of >1mm in 2 or more leads and/or T wave inversions in 2 or more contiguous leads.
   * Congenital long QT syndrome.
   * History of or presence of significant ventricular or atrial arrhythmia.
   * Clinically significant resting bradycardia (<50 beats per minute).
   * QTc >450 msec on screening ECG (using the QTcF formula).
   * Right bundle branch block plus left anterior hemiblock, bifascicular block.
   * Myocardial infarction within 3 months prior to starting Ponatinib.
   * Angina pectoris.
3. Other clinically significant vascular and heart disease (e.g., congestive heart failure, uncontrolled hypertension, history of labile hypertension, or history of poor compliance with an antihypertensive regimen).
4. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of Ponatinib (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
5. Uncontrolled hypertriglyceridemia (triglycerides >450 mg/dL).
6. Taking medications that are known to be associated with Torsades de Pointes and medications or herbal supplements that are known to be strong inhibitors of CYP3A4 within at least 14 days before the first dose of ponatinib.
7. History of or current autoimmune disease.
8. Systemic cancer chemotherapy within 2 weeks prior to study.
9. Known hypersensitivity to immunoglobulins or to any other component of the study drug formulation.
10. Active malignancy other than ALL with the exception of basal cell or squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix.
11. Active infection, any other concurrent disease or medical condition that are deemed to interfere with the conduct of the study as judged by the investigator.
12. Nursing women or women of childbearing potential not willing to use an effective form of contraception during participation in the study and at least 3 months thereafter or male patients not willing to ensure effective contraception during participation in the study and at least three months thereafter.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2021-09-08 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Number of patients who are event-free | at 5 months
  event-free survival rate

CONTACTS AND LOCATIONS:
Locations (15):
- Italy (15):
  - Area Vasta N. 5 Ascoli Piceno - S. Benedetto Del Tronto, Presidio Ospedaliero Av5 Osp. Gen. Prov.Le "C.G.Mazzoni" - Uoc Ematologia, Ascoli Piceno
  - Irccs Oncologico Istituto Tumori Giovanni Paolo Ii - Bari - Uo Ematologia, Bari
  - Asst Papa Giovanni Xxiii - Ospedale Di Bergamo - Sc Ematologia, Bergamo
  - As Dell'Alto Adige, Ospedale Centrale Di Bolzano - Ematologia E Centro Trapianto Midollo Osseo, Bolzano
  - Asst Degli Spedali Civili Di Brescia - Uo Ematologia, Brescia
  - Aulss 3 Serenissima, Ospedale Dell'Angelo - Mestre - Uo Ematologia, Mestre
  - Aou Di Modena - Sc Ematologia, Modena
  - Asl Salerno, Presidio Ospedaliero Tortora Pagani - Ematologia, Pagani
  - Ao Di Perugia, Ospedale S. Maria Della Misericordia - Ematologia E Trapianto Midollo Osseo, Perugia
  - Ao Ospedali Riuniti Marche Nord - Ospedale San Salvatore - Pesaro - Uoc Ematologia E Centro Trapianti, Pesaro
  - Asl Di Piacenza, Ospedale "Guglielmo Da Saliceto" - Ematologia E Centro Trapianti, Piacenza
  - Università Degli Studi Di Roma "Sapienza" - Dipartimento Di Medicina Traslazionale E Di Precisione - U.O.C. Ematologia, Roma
  - Ente Ecclesiastico Casa Sollievo Della Sofferenza - San Giovanni Rotondo - Ematologia, San Giovanni Rotondo
  - Aou Senese - Uoc Ematologia E Trapianti, Siena
  - Asui Di Udine - Presidio Ospedaliero "Santa Maria Della Misericordia" - Clinica Ematologica, Udine